CLINICAL TRIAL: NCT07378618
Title: Accuracy of Palatal Orthodontic Miniscrew Placement: Static vs Dynamic Computer-Guided Techniques in a Randomized Clinical Trial.
Brief Title: Evaluation of the Accuracy of Palatal Orthodontic Miniscrew Placement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, DDS, PhD, Associate Professor., University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS_StaticVsDynamic
Record Dates: First submitted 2026-01-13; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Malocclusion; Orthodontic Anchorage Procedures; Orthodontics
Keywords: miniscrews; computer guided surgery; TADs; orthodontics
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: This investigation is designed as an interventional, parallel-cohort randomized clinical study aimed at comparing two computer-assisted surgical approaches for palatal paramedian orthodontic miniscrew placement. Eligible participants are prospectively enrolled and are allocated in a 1:1 ratio to one of two parallel intervention cohorts: static computer-assisted surgery (s-CAS) or dynamic computer-assisted surgery (d-CAS). Randomization is performed at the participant level, and each subject receives only one type of intervention, with no crossover between cohorts.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static computer-guided surgery group (Active Comparator): Participants allocated to this arm undergo palatal paramedian orthodontic miniscrew placement using a static computer-assisted surgical protocol. Preoperative planning is performed by integrating cone-beam computed tomography (CBCT) data with intraoral digital scans to define the planned miniscrew position, trajectory, and insertion depth. Based on the virtual plan, a patient-specific stereolithographic surgical guide is digitally designed to adapt to the palatal anatomy and to extend to the posterior dentition in order to ensure stability.
  The surgical guide is fabricated using biocompatible resin through additive manufacturing and will be verified intraorally for proper fit prior to miniscrew insertion. Miniscrew placement is performed under local anesthesia using the static guide, which constrains the insertion path and depth according to the preoperative plan. Two self-drilling orthodontic miniscrews of standardized dimensions are placed in the paramedian palatal region.
  Interventions: Procedure: Computer-guided Miniscrew insertion
- Dynamic computer-guided surgery (Experimental): Participants allocated to this arm undergo palatal paramedian orthodontic miniscrew placement using a dynamic computer-assisted navigation system. Preoperative planning is conducted by merging CBCT datasets with intraoral digital scans within a dedicated navigation software environment to define the planned miniscrew position, angulation, and insertion depth. No physical surgical guide is produced for this intervention.
  Real-time navigation is enabled through the registration of a jaw reference tool and a handpiece tracking system, which allow continuous monitoring of instrument position relative to the patient's anatomy. Miniscrew insertion is performed under local anesthesia while the operator follows real-time visual feedback displayed on the navigation interface, enabling ongoing verification and, when necessary, intraoperative adjustment of the insertion trajectory.
  Two self-drilling orthodontic miniscrews of standardized dimensions are inserted in the paramedian palatal regio
  Interventions: Procedure: Computer-guided Miniscrew insertion

INTERVENTIONS:
Procedure: Computer-guided Miniscrew insertion — This intervention consists of a standardized digital workflow for orthodontic miniscrew placement in the paramedian region of the maxillary palate.
  Based on this integrated dataset, miniscrew position, angulation, and insertion depth are virtually planned to achieve bicortical anchorage while respecting predefined safety margins. Miniscrew insertion is performed under local anesthesia using self-drilling orthodontic miniscrews of standardized dimensions, without pre-drilling. Depending on group allocation, placement is carried out using either a static surgical guide or real-time dynamic navigation, while imaging acquisition and planning protocols remain identical. Immediate postoperative CBCT imaging is obtained to verify miniscrew position and to allow quantitative accuracy assessment.

SUMMARY:
This randomized clinical trial has the objective of comparing the accuracy of palatal paramedian miniscrew placement using static computer-assisted surgery (s-CAS) and dynamic computer-assisted surgery (d-CAS).

A population of forty subjects requiring palatal paramedian miniscrew insertion is going to be randomized into two groups to receive two miniscrews placed with s-CAS (Group A; n=20 subjects, 40 miniscrews) and d-CAS (Group B; n=20 subjects, 40 miniscrews). Preoperative digital intraoral scans and CBCT images will be used for virtual planning. Group A procedures is going to employ patient-specific surgical guides, while group B procedures is going to be performed with real-time navigation. Immediate postoperative CBCT scans will be superimposed to measure four accuracy parameters: coronal, apical, depth, and angular deviation from the planned position. Statistical analysis will include Student's t-test or Mann-Whitney U test as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* (1) subjects in late mixed dentition or permanent dentition,
* (2) a need for orthodontic or orthopedic treatment and no previous treatments,
* (3) good oral hygiene,
* (4) absence of acute infection in the oral cavity,
* (5) good general health

Exclusion Criteria:

* (1) syndromic patients
* (2) uncontrolled systemic diseases.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Apical deviation | Perioperative/Periprocedural
  The linear deviation at the apical endpoint of the miniscrew (in millimeters)
Coronal deviation | Perioperative/Periprocedural
  The linear deviation at the coronal entry point of the miniscrew (in millimeters)
Depth deviation | Perioperative/Periprocedural
  quantifies the vertical displacement of the apical tip (in millimeters)
angular deviation | Perioperative/Periprocedural
  the angular difference between the planned and actual screw trajectories (in angular degrees)

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, Roma, Italy

IPD SHARING:
Plan to Share IPD: No